CLINICAL TRIAL: NCT07291245
Title: Kawasaki MATCH: A Clinical Decision Support Tool to Detect KD
Brief Title: Kawasaki MATCH Trial
Acronym: MATCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Gordon and Marilyn Macklin Foundation (Unknown); Rady Children's Hospital, San Diego (Other)
Responsible Party: Principal Investigator, Michael Gardiner, Associate Clinical Professor, Associate Division Chief of Research, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 140220; 68060 (Other Grant/Funding Number: Gordon and Marilyn Macklin Foundation)
Record Dates: First submitted 2025-11-24; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Kawasaki Disease
Keywords: Kawasaki Disease; Machine-learning; Artificial Intelligence (AI); Decision support; Point-of-care
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kawasaki MATCH (Experimental): Providers encouraged to access and utilize the Kawasaki MATCH decision support tool when evaluating and managing patients in the Emergency Department
  Interventions: Other: Kawasaki MATCH
- Routine Care (No Intervention): Providers prompted to manage patients as per usual/routine care without additional decision support.

INTERVENTIONS:
Other: Kawasaki MATCH — Providers access the Kawasaki MATCH decision support tool. Patient information is entered into the tool and a risk score is indicated to the provider. Kawasaki MATCH is a previously validated machine-learning decision support tool for the diagnosis of Kawasaki Disease. This tool utilizes patient age, 18 laboratory features, and 5 clinical features to formulate a risk score.
  Arms: Kawasaki MATCH

SUMMARY:
Evaluating the impact of a machine-learning clinical decision support tool on provider practice when evaluating febrile patients with Kawasaki Disease (KD) and non-KD illnesses.

DETAILED DESCRIPTION:
Following laboratory evaluation, providers will be randomized to treat patients according to usual practice/standard of care vs. receiving clinical decision support from the Kawasaki MATCH tool - a previously validated machine-learning clinical decision support tool to identify Kawasaki Disease. The study aim is to evaluate the accuracy of Kawasaki MATCH prospectively when used at the point of care, as well as how this tool impacts clinical decisions including additional evaluation and hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* Measured or subjective fever for >= 3 calendar days
* One measured fever >= 38.0 C (home or in ED)
* One or more clinical feature of Kawasaki Disease including:
* Rash
* Conjunctival injection
* Oropharyngeal changes
* Extremity changes (erythema, edema, desquamation)
* Cervical adenopathy (>=1.5cm)
* Infants < 6 months of age with >= 7 days of fever eligible even if none of the above clinical features
* Requires IV/phlebotomy for clinical evaluation

Exclusion Criteria:

* Congenital or Acquired Immune function
* Genetic disorders
* Current systemic steroid, immunosuppression, or chemotherapy treatment (not including inhaled steroids)

Ages: 30 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Time to Kawasaki Disease treatment (KD patients only) | 90 days
  Time in days from initial ED evaluation to initial IVIG treatment in patients ultimately diagnosed with Kawasaki Disease

SECONDARY OUTCOMES:
Kawasaki MATCH score | Day 1 (day of enrollment)
  MATCH score determined by entering patient clinical and laboratory information into the Kawasaki MATCH algorithm. Algorithm output is a decimal between 0 and 1. Scores less than 0.4 will be deemed a prediction of "not Kawasaki Disease" while scores of 0.4 or higher will be deemed "Kawasaki Disease"
Hospital Admission Rate | Day 1 (day of enrollment)
  Proportion of patients admitted to the hospital from the Emergency Department (ED).
  Admitted patients = 1 Discharged patients = 0
Kawasaki Disease consultation rate | Day 1 (day of enrollment)
  Proportion of patients receiving Kawasaki service consultation
ED return visit | 7 days
  Return to Emergency Department
Additional interventions | Day 1 (day of enrollment)
  Additional ED orders for laboratory/imaging studies or additional procedures after the time of randomization
Provider assessment of KD likelihood - baseline | Day 1 (day of enrollment)
  Visual analog scale of suspected likelihood of Kawasaki Disease. Scale between 0 (Definitely not Kawasaki Disease) and 100 (Definitely Kawasaki Disease) with higher values indicating higher provider suspicion for Kawasaki Disease.
  This outcome will be assessed on providers randomized to both study arms
Provider assessment of KD likelihood - after algorithm | Day 1 (day of enrollment)
  Visual analog scale of suspected likelihood of Kawasaki Disease. Scale between 0 (Definitely not Kawasaki Disease) and 100 (Definitely Kawasaki Disease) with higher values indicating higher provider suspicion for Kawasaki Disease.
  This outcome only assessed for providers in the experimental arm.
Algorithm helpfulness | Day 1 (day of enrollment)
  Visual analog scale of the perceived helpfulness of the Kawasaki MATCH algorithm. Scale between 0 (Not helpful) and 100 (Extremely helpful) with higher values indicating increased helpfulness.
  This outcome only assessed for providers in the experimental arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Rady Children's Hospital, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Not included in consent documents

REFERENCES:
- [Background] Lam JY, Shimizu C, Gardiner MA, Giorgio T, Wright V, Baker A, Anderson MS, Heizer H, Mohandas S, Kazarians A, Kaneta K, Jone PN, Dominguez SR, Szmuszkovicz JR, Newburger JW, Tremoulet AH, Burns JC. External Validation of a Machine Learning Model to Diagnose Kawasaki Disease. J Pediatr. 2025 Jul;282:114543. doi: 10.1016/j.jpeds.2025.114543. Epub 2025 Mar 21. PMID 40122277
- [Background] Lam JY, Shimizu C, Tremoulet AH, Bainto E, Roberts SC, Sivilay N, Gardiner MA, Kanegaye JT, Hogan AH, Salazar JC, Mohandas S, Szmuszkovicz JR, Mahanta S, Dionne A, Newburger JW, Ansusinha E, DeBiasi RL, Hao S, Ling XB, Cohen HJ, Nemati S, Burns JC; Pediatric Emergency Medicine Kawasaki Disease Research Group; CHARMS Study Group. A machine-learning algorithm for diagnosis of multisystem inflammatory syndrome in children and Kawasaki disease in the USA: a retrospective model development and validation study. Lancet Digit Health. 2022 Oct;4(10):e717-e726. doi: 10.1016/S2589-7500(22)00149-2. PMID 36150781

DOCUMENTS (2):
  • Study Protocol (2025-08-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT07291245/Prot_000.pdf
  • Statistical Analysis Plan (2025-12-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT07291245/SAP_001.pdf